CLINICAL TRIAL: NCT00596960
Title: Motivating Chronic Hepatitis C Patients to Reduce Alcohol Use
Brief Title: Study of the Effects of Motivational Enhancement Therapy on Alcohol Use in Chronic Hepatitis C Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEUA-009-07S
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2014-11-28 (Estimated); Last update posted 2014-11-28 (Estimated); Status verified 2014-11

CONDITIONS: Alcohol Dependence; Chronic Hepatitis C
Keywords: Alcohol Abuse; Alcohol Dependence; Carbohydrate Deficient Transferrin; Drug Dependence; Hepatitis C; Motivation
MeSH Terms: conditions — Alcoholism; Hepatitis C, Chronic; Substance-Related Disorders; Hepatitis C | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Enhancement Therapy (Experimental): Motivational enhancement therapy
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)
- Health Education (Active Comparator): health education intervention
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy (MET) — MET is a 4 session intervention based on motivational approaches that was successful in project MATCH.
  Arms: Motivational Enhancement Therapy
Behavioral: Health education — Health education intervention will serve as the active control. The intervention will consist of 4 sessions of health education with a focus on sleep hygiene, nutrition, exercise and relaxation training.
  Arms: Health Education

SUMMARY:
The purpose of this study is to determine whether motivational enhancement therapy (MET) reduces alcohol use in a population of HCV-infected veterans who are currently drinking alcohol and have alcohol disorders. We hypothesize that veterans with HCV, an alcohol use disorder and continued excessive alcohol use who receive MET will have a greater reduction in the number of standard alcohol drinks per week and a greater percentage of days abstinent than veterans who receive health education control intervention.

DETAILED DESCRIPTION:
BACKGROUND: Recent studies suggest the presence of hepatitis C virus (HCV) among veterans treated within the Veterans Affairs Medical Center is 3 to 4 times more common than among the general population and approximately 50 to 60% of the patients are at risk for progression to end-stage liver disease. Alcohol use substantially increases the rate of liver disease progression. Alcohol treatment based on motivational principles has been found to be effective in alcohol treatment seeking individuals with low levels of psychiatric comorbidity. Effective treatments for alcohol use have not been studied in patients chronically infected with HCV, individuals who typically do not seek separate specialty care for alcohol problems. The primary purpose of this study is to determine the efficacy of motivational enhancement therapy (MET) in reducing alcohol use in a population of HCV-infected veterans who are currently drinking alcohol and have alcohol disorders. Secondarily this study is designed to determine whether changes in motivation predict changes in alcohol use; determine whether MET effects non-alcohol related behavior such as adherence to clinic appointments and the effects of a reduction in alcohol use on biomarkers of alcohol use and HCV viral load.

METHODS: Two sites of the national VA Hepatitis C Resource Center, including Minneapolis and Portland will enroll 136 men, women, and minority veterans who are HCV positive, have an alcohol use disorder and are currently drinking. Participants will be recruited from the hepatitis clinics at each site after they have received two sessions of care from hepatitis clinicians. Subjects will be eligible for enrollment in the study if they are drinking at least 7 drinks per week over the preceding 2-weeks. Participants will be randomly assigned to one of two groups: a 4-week session MET or a 4 session health education control intervention. Follow-up data will be collected at 3 and 6 month interviews by a blinded interviewer assessing current alcohol use. Secondary outcomes including stage of change, data regarding enrollment and attendance in separate substance abuse treatment or self-help programs (Alcoholics Anonymous) will be collected from participants' medical record. HCV viral titers will be obtained at baseline and 6-months. Percent CDT and ethyl glucuronide will be measured to confirm self-reported alcohol use at each study visit. The primary outcome (efficacy of MET in reducing alcohol use) data will be analyzed using mixed effect models if the data are normally distributed and generalized estimated equations if the data are non-normally distributed.

CLINICAL RELEVANCE: This study focuses on a current VHA priority: treatment of veterans with HCV. Alcohol use on this population is a major risk factor for progression of liver disease. We anticipate that the MET proposed in this study will result in a slowing of the progression of liver disease, improvement in physical health, and a reduction in long-term service utilization and mortality rates.

POTENTIAL IMPACT ON VETERANS HEALTH CARE: Effectively addressing alcohol use disorders in a hepatitis clinic will contribute to a new standard of care for HCV patients within VA. MET is a relatively brief, easily adaptable intervention that if effective is likely to improve access to alcohol treatment, acceptance by patients and improve clinical efficiency. In addition, reducing or eliminating alcohol use in this population has the potential to alter the course of liver disease progression, reducing the rates of cirrhosis, hepatocellular carcinoma and the need for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 or older
* Serum antibody and polymerase chain reaction positive for hepatitis C
* Drinking greater than 7 drinks for each of the proceeding 2 weeks or one day heavy drinking day per week for 2 week (heavy drinking day:>4 drinks in one day)
* Diagnosed with alcohol abuse or dependence

Exclusion Criteria:

* Diagnosis of cocaine, methamphetamine or opioid dependence within the past 6 months
* Unable to attend clinic appointments
* Any known pre-existing medical conditions that could interfere with participation in the protocol, such as: CNS trauma, known cognitive impairment, dementia, encephalopathy from liver disease, acute psychiatric instability, such as significant psychosis, mania, or elevated risk for suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-11; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric W. Dieperink, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - VA Medical Center, Portland, Portland, Oregon

REFERENCES:
- [Result] Dieperink E, Fuller B, Isenhart C, McMaken K, Lenox R, Pocha C, Thuras P, Hauser P. Efficacy of motivational enhancement therapy on alcohol use disorders in patients with chronic hepatitis C: a randomized controlled trial. Addiction. 2014 Nov;109(11):1869-77. doi: 10.1111/add.12679. Epub 2014 Aug 14. PMID 25040898

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Motivational enhancement therapy
  Motivational Enhancement Therapy (MET): MET is a 4 session intervention based on motivational approaches that was successful in project MATCH.
- Arm 2: health education intervention
  Health education: Health education intervention will serve as the active control. The intervention will consist of 4 sessions of health education with a focus on sleep hygiene, nutrition, exercise and relaxation training.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 70 | 69 (One subject did not have any alcohol use data and thus was excluded from the statistical analysis)
Completed | 59 | 60
Not Completed | 11 | 9
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Incarcerated | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — No alcohol use data | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 70 | 69 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (6.8) | 55.2 (6.3) | 55.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 68 | 65 | 133
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 48 | 46 | 94
  African American | 20 | 21 | 41
  Native American | 0 | 2 | 2
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 70 | 69 | 139
Percentage of days abstinent [Mean (Standard Deviation); unit: percentage of days abstinent] — Percentage of days abstinent from alcohol as measured by the time line follow back method in the past 30 days.
  percentage of days abstinent | 34.98 (26.7) | 34.63 (27.0) | 34.81 (26.8)
Mean standard drinks per week [Mean (Standard Deviation); unit: Standard drinks of alcohol] | 35.45 (25.42) | 38.86 (46.19) | 37.13 (37.03)
Beck Depression Inventory-II [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory-II is a continuous measure of depressive symptoms. Maximum score is 63 with a range of 0 to 63. Higher scores indicate more severe depressive symptoms.
  units on a scale | 17.40 (11.58) | 17.31 (10.79) | 17.36 (11.16)
Brief Symptom Inventory [Mean (Standard Deviation); unit: units on a scale] — The Brief Symptom Inventory (BSI) is a 53 item self-report instrument that reflects 9 symptom dimensions: Somatization (SOM), Obsessive-compulsive (0-C), Interpersonal sensitivity (I-S), Depression (DEP), Anxiety (ANX), Hostility (HOS), Phobic anxiety (PHOB), Paranoid ideation (PAR) and Psychotics (PSY). For this study we used a total BSI score as a measure of distress. The maximum score is 159 and a range of 0 to 159 with higher scores indicating more psychological distress.
  units on a scale | 51.23 (41.23) | 56.91 (44.18) | 54.05 (42.66)
Posttraumatic stress disorder checklist - Civilian (PCL-C) [Mean (Standard Deviation); unit: units on a scale] — The PCL-C is a standardized self-report rating scale for Posttraumatic Stress disorder symptoms (PTSD). The maximum score is 85 with a range of 17 to 85. Higher scores indicate increased PTSD symptoms. A cut-off of 50 has good sesnitivity and specificty for PTSD.
  units on a scale | 38.01 (15.21) | 40.61 (16.04) | 39.28 (15.62)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Alcohol Drinks Per Week (as Measured by the Time Line Follow Back Procedure) at the 6 Month Follow-up.
Description: A standard drink was considered 14 oz. of alcohol or12 oz of regular beer, 5 oz of regular wine, or 1.5 oz of distilled spirits. The number of drinks per week was measured for 30 a day time frame at baseline, 3 months and 6-months.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Standard Alcohol drinks
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 70 | 68
Standard Alcohol drinks | 14.88 (27.94) | 21.41 (29.39)

2. Primary Outcome: Percent Days Abstinent From Alcohol at 6 Months
Description: Alcohol use was measured for 30 days at baseline, 3-months and 6-months using the time-line follow back method. Percent days abstinent was measured by determining: days abstinent/30days X 100=%days abstinent.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 70 | 68
percentage of days abstinent | 73.15 (32.18) | 59.49 (35.30)

3. Secondary Outcome: Heavy Drinking Days (Greater or Equal to 4 Drinks)
Description: This was measured as heavy drinking days per 30 day time frame. A standard drink was considered 14 oz. of alcohol or12 oz of regular beer, 5 oz of regular wine, or 1.5 oz of distilled spirits. A heavy drinking day was considered to be 4 or greater drinks during a day.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: heavy drinking days
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 70 | 68
heavy drinking days | 5.10 (8.1) | 7.38 (9.53)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 7/70 | 14/69
Other Adverse Events (participants affected / at risk) | 0/70 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=70) | Arm 2 (N=69)
Liver failure (Hepatobiliary disorders) | 1 (1) | 3 (3) — Death
psychiatric symptoms (Psychiatric disorders) | 1 (1) | 2 (2) — hospitalization
Alcohol intoxication (Psychiatric disorders) | 2 (2) | 4 (4) — Hospitalization
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — Death
GI distress (Hepatobiliary disorders) | 1 (1) | 3 (3) — Hospitalization
fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — hospitalization
chest pain (Cardiac disorders) | 0 (0) | 1 (1) — Hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes